CLINICAL TRIAL: NCT00598026
Title: Evaluation of the " Tele-follow-up " for the Follow-up of Implantable Defibrillators
Acronym: EVATEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35RC07_9901; 0203/076 (Other: Internal (CIC)); 2007-A00888-45 (Other: IDRCB); LOC/07-04 (Other: Former internal Identifier)
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Defibrillators, Implantable; Telemedicine
Keywords: Tele medicine; ICD follow-up; Cost / benefit study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tele- follow-up: remote transmission to the implantation centre every 3 months
  Interventions: Other: Tele- follow-up
- 2 (Active Comparator): Conventional follow-up: visits at the implantation centre every 3 months
  Interventions: Other: Conventional follow-up

INTERVENTIONS:
Other: Tele- follow-up — Remote transmission to the implantation centre every 3 months
  Arms: 1
Other: Conventional follow-up — Visits at the implantation centre every 3 months
  Arms: 2

SUMMARY:
The implantable cardioverter defibrillator (ICD) has been shown to be effective in preventing mortality in patients with ventricular tachyarrhythmia. However, the expanding indications of this therapy will have an impact on the follow-up policy. Currently, regular follow-up visits are scheduled every 3 months. In this context, the recently-introduced "remote monitoring" devices constitute a promising new technique, allowing to transmit information about the status of the device and ICD therapies, without direct contact between patients and physicians. This monitoring by "tele-follow-up" might reduce the cost of care by avoiding useless visits to the implantation centre.

The aim of our study is to assess the cost-benefit ratio of "tele-follow-up" assisted care as compared with the conventional ICD follow-up.

DETAILED DESCRIPTION:
The implantable cardioverter defibrillator (ICD) has been shown to be effective in preventing mortality in patients with ventricular tachyarrhythmia. However, the expanding indications of this therapy will have an impact on the follow-up policy. Currently, regular follow-up visits are scheduled every 3 months. In this context, the recently-introduced "remote monitoring" devices constitute a promising new technique, allowing to transmit information about the status of the device and ICD therapies, without direct contact between patients and physicians. This monitoring by "tele-follow-up" might reduce the cost of care by avoiding useless visits to the implantation centre.

The aim of our study is to assess the cost-benefit ratio of "tele-follow-up" assisted care as compared with the conventional ICD follow-up. Thanks to an open label, randomized, 2 arms study : one using a telephone follow up, the other a conventional follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18,
* First implantation of an implantable cardioverter defibrillator device (CRT-D devices being excluded), single or dual-chamber in primary or secondary prevention,
* ICD with data-transmission features,
* GSM mobile phone network at patient home compatible with remote transmission,
* Patient able to use correctly the transmission system,
* Patients having given a written informed consent.

Exclusion Criteria:

* Class IV of NYHA,
* Concomitant pathology leading to a life expectancy inferior to the protocol duration,
* Concomitant participation to another protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1501 (Actual)
Dates: Start 2008-01-14 (Actual); Primary Completion 2011-03-07 (Actual); Study Completion 2011-03-07 (Actual)

PRIMARY OUTCOMES:
Rate of major cardiovascular events: all cause death, hospitalisation for a cardiovascular event, unsuccessful ICD therapies, and inappropriate ICD therapies. | 1 year

SECONDARY OUTCOMES:
Time to onset of the first major cardiovascular event (censored criterion) | 1 year
Death rate | 1 year
Hospitalisation rate for a cardiovascular event | 1 year
Rate of unsuccessful or inappropriate ICD therapies | 1 year
Mean costs of each follow-up strategy | 1 year
Number of non programmed additional consultations at the implantation centre | 1 year
Number and cause of device re-programming | 1 year
Number of drop-outs in the tele-follow-up group | 1 year
Adherence of the patients to the tele-follow-up strategy | 1 year
Feasibility of the tele-follow-up in implantation centres | 1 year
Cost-benefit analysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe MABO, MD, PhD, Study Director — Rennes University Hospital; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital; Isabelle DURAND-ZALESKI, MD, PhD, Study Chair — Creteil University Hospital
Locations (30):
- France (30):
  - Service de Cardiologie - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Service de Cardiologie - CHU d'Angers, Angers
  - Service de Cardiologie - CHU Jean Minjoz, Besançon
  - Service de Cardiologie -Hôpital de la Cavale Blanche, Brest
  - Service de Cardiologie - Groupement Hospitalier Est de Lyon, Bron
  - Service de Cardiologie - Hôpital de la Côte de Nacre, Caen
  - Service de Cardiologie - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Service de Cardiologie - Hôpital Henri Mondor, Créteil
  - Centre de Cardiologie - CHU de Dijon, Dijon
  - Service de cardiologie et Urgences cardiologiques - Hôpital Michallon, Grenoble
  - Cardiologie A - CHRU de Lille, Lille
  - Service de Cardiologie - CHU de Limoges, Limoges
  - Service de Cardiologie - CHU Timone Adultes, Marseille
  - Département de Cardiologie - CHU de Montpellier, Montpellier
  - Service de Cardiologie - Institut du Thorax - Hôpital Laennec, Nantes
  - Service de Cardiologie - Hôpital Pasteur, Nice
  - Service de Cardiologie - CHU de Nîmes, Nîmes
  - Service de Cardiologie - Hôpital Européen Georges Pompidou, Paris
  - Service de Cardiologie - Hôpital Lariboisière, Paris
  - Institut de Cardiologie - Hôpital de la Pitité Salpétrière, Paris
  - Hôpital Cardiologique du Haut Lévêque - CHU de Bordeaux, Pessac
  - Service médico-chirurgical de Cardiologie - CHU de Poitiers, Poitiers
  - Département de Cardiologie - CHU de Reims, Reims
  - Département de Cardiologie et Maladies Vasculaires - Hôpital de Pontchaillou, Rennes
  - Service de Cardiologie - Hôpital Charles Nicolle, Rouen
  - Service de Cardiologie - CHU de Saint Etienne, Saint-Etienne
  - Service de Cardiologie - Hôpital de Hautepierre, Strasbourg
  - Service de Chirurgie Cardiovasculaire - Hôpital Rangueil, Toulouse
  - Service de Cardiologie B - Hôpital Trousseau, Tours
  - Département de Cardiologie - CHU de Nancy-Brabois, Vandœuvre-lès-Nancy